CLINICAL TRIAL: NCT03663439
Title: Evaluation of Modified Shell Technique Versus Onlay Bone Graft for Reconstruction of Atrophic Anterior Maxilla
Brief Title: Modified Shell Technique Versus Onlay Bone Graft in Anterior Maxilla
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr hisham mohamed, Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1552016
Record Dates: First submitted 2018-09-05; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Implant Complication
Keywords: anterior augmentation,shell technique,onlay bone graft

STUDY DESIGN:
Intervention Model Description: control group (modified shell technique) study group (onlay bone graft)
Who Masked: Outcomes Assessor
Masking Description: control group (modified shell technique) study group (onlay bone graft)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified shell technique (Experimental): block of bone from the mandibular ramus divided into two shells ,grafting one shell in the anterior maxilla to increase width
  Interventions: Procedure: modified shell technique
- onlay bone graft (Active Comparator): grafting block of bone from the mandibular ramus in the atrophic anterior maxilla
  Interventions: Procedure: modified shell technique

INTERVENTIONS:
Procedure: modified shell technique — divided block of bone into two shells and grafting one shell in anterior maxilla

SUMMARY:
Amount of bone volume and (width and height):

Will be measured using linear measurements from CBCT after 6 month from implant insertion.

Will be measured using Histometric analysis of bone area percent sampling from recipient site after 6 months.

DETAILED DESCRIPTION:
Augmentation of insufficient bone volume can be brought about by different methods, including, particulate and block grafting materials, Guided Bone Regeneration with or without growth and differentiation factors, ridge splitting, expansion and distraction osteogenesis, either alone or in combination. These techniques may be used for horizontal/vertical ridge augmentation

Autograft is considered as the Gold Standard for bone transplantation and various studies have shown efficacy for it. It is osteogenic, osteoconductive and osteoinductive. Autografts can be derived from extra oral source (iliac crest, ribs) or intraoral source (chin, ramus). They can be used in block or particulate form. Corticocancellous block grafts are preferred because of enhanced revascularization of the cancellous portion, and mechanical support and rigidity of the cortical portion, which ensures optimal ridge augmentation.

Fouad Khoury presented a three-dimensional (3D) reconstruction technique for atrophic ridges and complicated vertical bone defects using mandibular bone block graft "the Gold standard". There are several possibilities for augmentation of bone volume depending on situation, indication and adequate diagnosis; the treatment options can be extended from minimally invasive procedures with locally harvested bone grafts in local anesthesia, to very sophisticated grafting techniques for 3D bone reconstruction with extra oral harvested bone grafts. Khoury reported that his ascending ramus grafts is almost 5 times more than chin grafts

ELIGIBILITY:
Inclusion Criteria:

* patients with atrophic anterior maxilla
* No intraoral soft and hard tissue pathology
* No systemic condition that contraindicate implant placement
* Both sexes.

Exclusion Criteria:

* Heavy smokers more than 20 cigarettes per day.
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems
* Immunodeficiency pathology, bruxism, stress situation (socially or professionally), emotional instability, and unrealistic aesthetic demands.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2018-09-16 (Estimated); Primary Completion 2018-09-20 (Estimated); Study Completion 2019-02-16 (Estimated)

PRIMARY OUTCOMES:
Histomorphometric | 3 months
  Type of bone formed by graft, after 3 months biopsy from the bone formed